CLINICAL TRIAL: NCT01823575
Title: Comparison of the Efficacy of Silicone-covered Metallic Ureteral Stent and Double-J Stent for Malignant Ureteral Obstruction: A Prospective Randomized Controlled Trial Based on Exploratory Research
Brief Title: Comparison of Silicone-covered Metallic Ureteral Stent and Double-J Stent for Malignant Ureteral Obstruction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hoon Shin, Associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JHS_URST
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Malignant Ureteral Obstruction
Keywords: malignant ureteral obstruction; silicone-covered metallic ureteral stent; double-J stent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silicone-covered metallic ureteral stent (Experimental): Deployment of a silicone-covered metallic ureteral stent for malignant ureteral obstruction and compare the results with placement of a double-J stent in terms of primary patency rate at 3 month follow-up (primary end point)
  Interventions: Device: Silicone-covered metallic stent
- Double-J stent (Active Comparator): Placement of a double-J stent for malignant ureteral obstruction and compare these results to deployment of a silicone-covered metallic stent in terms of primary patency rate at 3 month follow-up.
  Interventions: Device: Double-J stent

INTERVENTIONS:
Device: Silicone-covered metallic stent — deployment of silicone-covered metallic stent for malignant ureteral obstruction as a new therapy as compared with placement of double-J stent as a conventional therapy
  Arms: Silicone-covered metallic ureteral stent
Device: Double-J stent — Placement of double-J stent as a conventional treatment to be compared with a new experimental treatment - deployment of silicone-covered metallic stent
  Arms: Double-J stent

SUMMARY:
Malignant ureteral obstruction often necessitates chronic urinary diversion and is associated with high rates of failure with traditional double-J ureteral stents. To overcome drawbacks of the double-J stent, recently, metallic stents have been used to manage for palliative treatment in patients with ureteral obstruction associated with end stage malignant disease. The success rates of metallic stents have been reported to be high and the method proved to be useful in patients with malignant ureteral obstruction. In addition, covered metallic stents have many advantages compared with bare metallic stents, such as lower rate of tissue invasion and higher patency rate. However, there is little investigation about comparison of clinical efficacy between covered-metallic stents and double-J stents in malignant ureteral obstruction.

Therefore, investigators plan to perform a prospective randomized study to compare clinical efficacy of silicone-covered metallic ureteral stent and double-J ureteral stent in patients with malignant ureteral obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-80 years
2. Malignant mid- to distal ureteral obstruction by abdominal or pelvic malignancy with overt hydronephrosis documented on CT scans
3. Expected life expectancy more than three months

Exclusion Criteria:

1. History of unilateral nephrectomy or bladder reconstruction
2. History of kidney transplantation
3. History of severe allergy to contrast media
4. State of dialysis
5. Performance status - 3 or 4 on ECOG scale

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-08 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
primary patency rate at 3-month F.U. | 3 month after stent deployment
  Confirmation of patency of the stents with USG and renal biochemistry, without additional intervention.

SECONDARY OUTCOMES:
Primary patency rate at 6- and 12-month F.U. | at 6 and 12 months after stent deployment
  Confirmation of patency of the stents with USG and renal biochemistry, without additional intervention.
  Assessment of complications in two study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hoon Shin, M.D., Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea